CLINICAL TRIAL: NCT02079506
Title: An Open-label, Multiple-dosing, Two-arm, One-sequence, Crossover Study to Evaluate the Safety and Pharmacokinetics After Oral Concurrent Administration of Candesartan 32 mg and Rosuvastatin 20 mg in Healthy Male Volunteers
Brief Title: Pharmacokinetic Drug Interaction Between Candesartan and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DP-CTR208-I-01
Record Dates: First submitted 2014-03-04; First posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
MeSH Terms: interventions — candesartan; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental)
  Interventions: Drug: Candesartan
- Treatment B (Experimental)
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Candesartan
  Arms: Treatment A
Drug: Rosuvastatin
  Arms: Treatment B

SUMMARY:
The objective of this study is to compare pharmacokinetics after single oral administration of candesartan and rosuvastatin each separately versus coadministration of candesartan and rosuvastatin in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers af aged between 20 years to 45 years
* Have a weight above 55kg and Ideal body weight (IBW) between -20% and +20% inclusive
* Eligible subjects with acceptable medical history and physical examination

Exclusion Criteria:

- Have a known hypersensitivity or history of clinically significant hypersensitivity to drugs including the same class drugs with candesartan or rosuvastatin, or other drugs

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss of candesartan | 22 points
  0h(pre-dose), 1, 2, 3, 4, 5, 6, 7, 8, 12 and 24 h
Cmax,ss of candesartan | 22 points
  0h(pre-dose), 1, 2, 3, 4, 5, 6, 7, 8, 12 and 24 h
AUCτ,ss of rosuvastatin | 28 points
  0(pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 9, 12 and 24 h
Cmax,ss of rosuvastatin | 28 points
  0(pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 9, 12 and 24 h

SECONDARY OUTCOMES:
tmax,ss of candesartan | 22 points
  0h(pre-dose), 1, 2, 3, 4, 5, 6, 7, 8, 12 and 24 h
CLss/F of candesartan | 22 points
  0h(pre-dose), 1, 2, 3, 4, 5, 6, 7, 8, 12 and 24 h
Cmin,ss of candesartan | 22 points
  0h(pre-dose), 1, 2, 3, 4, 5, 6, 7, 8, 12 and 24 h
tmax,ss of rosuvastatin | 28 points
  0h(pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 9, 12 and 24 h
CLss/F of rosuvastatin | 28 points
  0h(pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 9, 12 and 24 h
Cmin,ss of rosuvastatin | 28 points
  0h(pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 9, 12 and 24 h

CONTACTS AND LOCATIONS:
Overall Officials: JangHee Hong, PhD., Principal Investigator — Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, Jung-gu, Daejeon, South Korea